CLINICAL TRIAL: NCT03131349
Title: Zinc and Iron in Children With Short Stature
Acronym: zincandiron
Status: Completed | Type: Observational
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, engy dawood, doctor, Assiut University
Other Study IDs: assiut university17100104
Record Dates: First submitted 2017-04-23; First posted 2017-04-27 (Actual); Last update posted 2020-10-30 (Actual); Status verified 2020-10

CONDITIONS: Zinc; Deficiency With Anemia

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 6 Months
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- column heading in tables: history examinations investigation:serum zinc and iron
  Interventions: Diagnostic Test: serum zinc and iron
- row heading in tables: history examinations investigation:serum zinc and iron
  Interventions: Diagnostic Test: serum zinc and iron

INTERVENTIONS:
Diagnostic Test: serum zinc and iron — history ,examination,investigations

SUMMARY:
Short stature is defined as height below 3rd centile or less than two standard deviations below the median height for that age and sex according to the population standard zinc and iron have important role in growth for children

DETAILED DESCRIPTION:
Short stature is defined as height below 3rd centile or less than two standard deviations below the median height for that age and sex according to the population standard.

Approximately 3% children in any population will be short, amongst which half will be physiological (familial or constitutional) and half will be pathological.

It is estimated that approximately 60%-80% of all short children at or below 2standerd deviation fit the definition of idiopathic short stature.

The growth and development of human require an adequate supply of many different nutritional factors. Nutritional deficiencies causing short stature include: those associated with stunting as: protein and zinc, nutrient associated with rickts as :vitamin D, and those with bone abnormalities as: cupper,zin,and vitamin c Insufficient nutrition tends to lead to short stature with a delayed pattern of growth. Under-nutrition can be isolated (eg, caused by inadequate food supply or self-imposed restriction, such as fear of obesity), or it may be a component of an underlying systemic disease that interferes with food intake or absorption, or increases energy needs. The hallmark of under-nutrition is low weight-for-height .

Trace elements are dietary mineral that are present in very minute quantities (less than 0.01%),they divided into three groups (WHO classification): Essential elements such as iodine and zinc ,Probably essential elements such as manganese and silicon , Potentially toxic elements such as fluoride,lead,cadmium, mercury, & Lithium.

Trace elements play significant functions as growth,oregulation of gene expression, immunity,the endocrine system, brain development, and the cell protection system. An adequate micronutrient intake is crucial for health, particularly in infants, children and adolescents ,deficiency in micronutrients can affect growth and development, particularly during periods of rapid growth.

ELIGIBILITY:
Inclusion Criteria:

* • children of both sexes.

  * Age range: 4-18 years.
  * patients fulfilling criteria of short stature.
* height is 2 standard deviations below normal .
* initial height below the third percentile on Egyptian growth chart. • Number of patients: will include 50 cases

Exclusion Criteria:

* Skeletal dysplasia.
* Chromosomal anomalies

Ages: 2 Years to 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: 50 cases will be included :35 child with idiopathic short stature and 25 as controls aging from4-18 years old coming to endocrinology clinic at Assuit University Children Hospital will be investigated for serum of zinc and iron
Sampling Method: Probability Sample
Enrollment: 50 (Actual)
Dates: Start 2017-06-01 (Actual); Primary Completion 2018-01-01 (Actual); Study Completion 2019-08-15 (Actual)

PRIMARY OUTCOMES:
zinc and iron in children with idiopathic short stature | 6 months
  Assessment of the serum level of zinc and iron in idiopathic with short stature.

CONTACTS AND LOCATIONS:
Locations (1):
- Engy dawood, Asiut, Egypt

IPD SHARING:
Plan to Share IPD: Undecided
patients aging 2-18years old will be dbtained at the start of the study